CLINICAL TRIAL: NCT02560428
Title: Evaluating System Change to Advance Learning and Take Evidence to Scale (ESCALATES)
Acronym: ESCALATES
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Texas (Other); Rutgers University (Other); HealthPartners Institute (Other); University of Michigan (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Deborah Cohen, Associate Professor, Oregon Health and Science University
Other Study IDs: 11482
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Program Evaluation
Keywords: Mixed Methods; Cardiovascular Health; Implementation Evaluation; Cardiovascular Prevention Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: ESCALATES — The investigators collect and analyze qualitative data to identify the most effective combinations of intervention strategies for various practice types, contexts, and organizational characteristics, and to understand why and how those combinations are effective. The investigators also gather de-identified quantitative data that the R18s collected.
  Other Names: EvidenceNOW

SUMMARY:
The purpose of this study is to evaluate approximately eight grants that will test interventions to improve cardiovascular disease prevention. The investigators will collect and analyze qualitative data to identify the most effective combinations of intervention strategies. The investigators will observe grantees and selected practices to understand why and how those combinations are effective. The investigators will also gather data from the grantees to assess how effective the interventions are.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate approximately eight different R18 grants that will test practice change interventions to improve cardiovascular disease (CVD) prevention screening. The investigators will collect and analyze quantitative data (context, process, and outcomes) to identify the most effective combinations of intervention strategies for various practice types in relation to practice structure, context, and organizational characteristics associated with change in outcomes. The investigators will collect qualitative data (observation, interviews, online diaries) from grantees and selected practices to understand why and how those combinations are effective. The investigators will also gather documents and de-identified quantitative data from grantees.

Evidence clearly shows that many people do not receive guideline-concordant health care; this is true even for low cost treatments such as Aspirin prescribing, Blood pressure and Cholesterol control and Smoking cessation (the ABCS) known to prevent cardiovascular disease (CVD). In hospitals and integrated care systems with substantial resources, large quality improvement campaigns have been shown to increase adherence to guidelines by creating communities of learning that change behavior on a large scale. Agency for Healthcare Research and Quality (AHRQ) and the Patient Centered Outcomes Research Institute (PCORI) are partnering to launch a campaign to promote the improvement of guideline-based CVD preventive care in small primary care practices with limited resources and experience with quality improvement ("Implementation" RFA-HS-14-008). The practices for each of these R18 grants will be in a contiguous geographic region. This study will evaluate each of these R18 implementation grants.

The investigators' strategy is to conduct a prospective observational analysis to evaluate the effectiveness of the R18s ABCS quality improvement initiatives. To do this, the investigators will collect and analyze qualitative data to identify the most effective combinations of intervention strategies for various practice types, contexts, and organizational characteristics, and to understand why and how those combinations are effective. The investigators will also gather de-identified quantitative data that the R18s collected.

ELIGIBILITY:
Inclusion Criteria:

* All R18 grant awardees are included in the study.

Exclusion Criteria:

* N/A

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all R18 grantees
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with AMI, coronary artery bypass graft, PCI or IVD, and who had documentation of used of aspirin or another antithrombotic during the measurement period. | Quarterly for 4 years
  Acute myocardial infarction (AMI), ischemic vascular disease (IVD), percutaneous coronary interventions (PCI)
Percentage of participants with diagnosis of hypertension and whose blood pressure was adequately controlled (<140/90 mmHg) during the measurement period. | Quarterly for 4 years
  Patients 18years and older and 85years or younger with at least one face to face visit and active diagnosis of essential hypertension at any time before the first date of month 7 of the measurement period and who did not (i) have an active diagnosis of pregnancy at any time during the measurement period; or (ii) have evidence of end stage renal disease, dialysis, or renal transplant before or during the measurement period
Percentage of participants considered at high risk of cardiovascular events who were prescribed or were on a statin therapy during the measurement period. | Quarterly for 4 years
  Patients 21 and older with at least one face to face visit who have an active diagnosis of clinical atherosclerotic cardiovascular, LDL-C result >= 190mg/dL, aged 40 to 75years at the beginning of the measurement period with an active diagnosis of diabetes with the highest LDL-C result of 70 to 189mg/ dL and who (i) did not have adverse effect, allergy or intolerance to statin medication therapy; (ii) did not have an active diagnosis of pregnancy or breastfeeding; (iii) did not receive palliative care; (iv) did not have an active liver disease or hepatic disease of insufficiency; (v) did not have end stage renal disease; or (vi) did not have a most recent LDL-C results<70mg/dL for patients with a diabetes diagnosis who are not currently receiving statin medication therapy during the current measurement period or any time period.
Percentage of participants who were screened for tobacco use and received cessation counseling intervention if identified as a tobacco user. | Quarterly for 4 years
  Patients 18years and older as of the first day of the measurement period with at least two visits during the measurement period

SECONDARY OUTCOMES:
Practice capacity for change measured by adaptive reserve (AR) | Baseline, immediately after intervention, 6 months post-intervention (4 years maximum)
Practice capacity for quality improvement measured by CPCQ | Baseline, immediately after intervention, 6 months post-intervention (4 years maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Cohen, PhD, Principal Investigator — OHSU, Department of Family Medicine

REFERENCES:
- [Background] Cohen DJ, Balasubramanian BA, Gordon L, Marino M, Ono S, Solberg LI, Crabtree BF, Stange KC, Davis M, Miller WL, Damschroder LJ, McConnell KJ, Creswell J. A national evaluation of a dissemination and implementation initiative to enhance primary care practice capacity and improve cardiovascular disease care: the ESCALATES study protocol. Implement Sci. 2016 Jun 29;11(1):86. doi: 10.1186/s13012-016-0449-8. PMID 27358078
- [Background] Weiner BJ, Pignone MP, DuBard CA, Lefebvre A, Suttie JL, Freburger JK, Cykert S. Advancing heart health in North Carolina primary care: the Heart Health NOW study protocol. Implement Sci. 2015 Nov 14;10:160. doi: 10.1186/s13012-015-0348-4. PMID 26577091
- [Background] Shelley DR, Ogedegbe G, Anane S, Wu WY, Goldfeld K, Gold HT, Kaplan S, Berry C. Testing the use of practice facilitation in a cluster randomized stepped-wedge design trial to improve adherence to cardiovascular disease prevention guidelines: HealthyHearts NYC. Implement Sci. 2016 Jul 4;11(1):88. doi: 10.1186/s13012-016-0450-2. PMID 27377404
- [Background] Kaufman A, Rhyne RL, Anastasoff J, Ronquillo F, Nixon M, Mishra S, Poola C, Page-Reeves J, Nkouaga C, Cordova C, Larson RS. Health Extension and Clinical and Translational Science: An Innovative Strategy for Community Engagement. J Am Board Fam Med. 2017 Jan 2;30(1):94-99. doi: 10.3122/jabfm.2017.01.160119. PMID 28062823
- [Background] Reck J. Primary care provider burnout: implications for states & strategies for mitigation. National Academy for State Health Policy. 2017 Jan.
- [Background] Solberg LI. What do we know and need to know about transforming primary care? Fam Pract. 2017 Aug 1;34(4):371-372. doi: 10.1093/fampra/cmx031. No abstract available. PMID 28475721
- [Background] Parchman ML, Fagnan LJ, Dorr DA, Evans P, Cook AJ, Penfold RB, Hsu C, Cheadle A, Baldwin LM, Tuzzio L. Study protocol for "Healthy Hearts Northwest": a 2 x 2 randomized factorial trial to build quality improvement capacity in primary care. Implement Sci. 2016 Oct 13;11(1):138. doi: 10.1186/s13012-016-0502-7. PMID 27737719
- [Background] Solberg LI, Kuzel A, Parchman ML, Shelley DR, Dickinson WP, Walunas TL, Nguyen AM, Fagnan LJ, Cykert S, Cohen DJ, Balasubramanaian BA, Fernald D, Gordon L, Kho A, Krist A, Miller W, Berry C, Duffy D, Nagykaldi Z. A Taxonomy for External Support for Practice Transformation. J Am Board Fam Med. 2021 Jan-Feb;34(1):32-39. doi: 10.3122/jabfm.2021.01.200225. PMID 33452080
- [Result] Sweeney SM, Hall JD, Ono SS, Gordon L, Cameron D, Hemler J, Solberg LI, Crabtree BF, Cohen DJ. Recruiting Practices for Change Initiatives Is Hard: Findings From EvidenceNOW. Am J Med Qual. 2018 May/Jun;33(3):246-252. doi: 10.1177/1062860617728791. Epub 2017 Sep 4. PMID 28868889
- [Result] Ono SS, Crabtree BF, Hemler JR, Balasubramanian BA, Edwards ST, Green LA, Kaufman A, Solberg LI, Miller WL, Woodson TT, Sweeney SM, Cohen DJ. Taking Innovation To Scale In Primary Care Practices: The Functions Of Health Care Extension. Health Aff (Millwood). 2018 Feb;37(2):222-230. doi: 10.1377/hlthaff.2017.1100. PMID 29401016
- [Result] Dorr DA, Cohen DJ, Adler-Milstein J. Data-Driven Diffusion Of Innovations: Successes And Challenges In 3 Large-Scale Innovative Delivery Models. Health Aff (Millwood). 2018 Feb;37(2):257-265. doi: 10.1377/hlthaff.2017.1133. PMID 29401031
- [Result] Hemler JR, Hall JD, Cholan RA, Crabtree BF, Damschroder LJ, Solberg LI, Ono SS, Cohen DJ. Practice Facilitator Strategies for Addressing Electronic Health Record Data Challenges for Quality Improvement: EvidenceNOW. J Am Board Fam Med. 2018 May-Jun;31(3):398-409. doi: 10.3122/jabfm.2018.03.170274. PMID 29743223
- [Result] Balasubramanian BA, Marino M, Cohen DJ, Ward RL, Preston A, Springer RJ, Lindner SR, Edwards S, McConnell KJ, Crabtree BF, Miller WL, Stange KC, Solberg LI. Use of Quality Improvement Strategies Among Small to Medium-Size US Primary Care Practices. Ann Fam Med. 2018 Apr;16(Suppl 1):S35-S43. doi: 10.1370/afm.2172. PMID 29632224
- [Result] Cohen DJ, Dorr DA, Knierim K, DuBard CA, Hemler JR, Hall JD, Marino M, Solberg LI, McConnell KJ, Nichols LM, Nease DE Jr, Edwards ST, Wu WY, Pham-Singer H, Kho AN, Phillips RL Jr, Rasmussen LV, Duffy FD, Balasubramanian BA. Primary Care Practices' Abilities And Challenges In Using Electronic Health Record Data For Quality Improvement. Health Aff (Millwood). 2018 Apr;37(4):635-643. doi: 10.1377/hlthaff.2017.1254. PMID 29608365
- [Result] Edwards ST, Marino M, Balasubramanian BA, Solberg LI, Valenzuela S, Springer R, Stange KC, Miller WL, Kottke TE, Perry CK, Ono S, Cohen DJ. Burnout Among Physicians, Advanced Practice Clinicians and Staff in Smaller Primary Care Practices. J Gen Intern Med. 2018 Dec;33(12):2138-2146. doi: 10.1007/s11606-018-4679-0. Epub 2018 Oct 1. PMID 30276654
- [Result] Perry CK, Damschroder LJ, Hemler JR, Woodson TT, Ono SS, Cohen DJ. Specifying and comparing implementation strategies across seven large implementation interventions: a practical application of theory. Implement Sci. 2019 Mar 21;14(1):32. doi: 10.1186/s13012-019-0876-4. PMID 30898133
- [Result] Baron AN, Hemler JR, Sweeney SM, Tate Woodson T, Cuthel A, Crabtree BF, Cohen DJ. Effects of Practice Turnover on Primary Care Quality Improvement Implementation. Am J Med Qual. 2020 Jan/Feb;35(1):16-22. doi: 10.1177/1062860619844001. Epub 2019 Apr 29. PMID 31030525
- [Result] Lindner S, Solberg LI, Miller WL, Balasubramanian BA, Marino M, McConnell KJ, Edwards ST, Stange KC, Springer RJ, Cohen DJ. Does Ownership Make a Difference in Primary Care Practice? J Am Board Fam Med. 2019 May-Jun;32(3):398-407. doi: 10.3122/jabfm.2019.03.180271. PMID 31068404
- [Result] Phillips RL Jr, Cohen DJ, Kaufman A, Dickinson WP, Cykert S. Facilitating Practice Transformation in Frontline Health Care. Ann Fam Med. 2019 Aug 12;17(Suppl 1):S2-S5. doi: 10.1370/afm.2439. No abstract available. PMID 31405869
- [Result] Sweeney SM, Hemler JR, Baron AN, Woodson TT, Ono SS, Gordon L, Crabtree BF, Cohen DJ. Dedicated Workforce Required to Support Large-Scale Practice Improvement. J Am Board Fam Med. 2020 Mar-Apr;33(2):230-239. doi: 10.3122/jabfm.2020.02.190261. PMID 32179606
- [Result] Cohen DJ, Sweeney SM, Miller WL, Hall JD, Miech EJ, Springer RJ, Balasubramanian BA, Damschroder L, Marino M. Improving Smoking and Blood Pressure Outcomes: The Interplay Between Operational Changes and Local Context. Ann Fam Med. 2021 May-Jun;19(3):240-248. doi: 10.1370/afm.2668. PMID 34180844
- [Result] Edwards ST, Marino M, Solberg LI, Damschroder L, Stange KC, Kottke TE, Balasubramanian BA, Springer R, Perry CK, Cohen DJ. Cultural And Structural Features Of Zero-Burnout Primary Care Practices. Health Aff (Millwood). 2021 Jun;40(6):928-936. doi: 10.1377/hlthaff.2020.02391. PMID 34097508
- [Result] Marino M, Solberg L, Springer R, McConnell KJ, Lindner S, Ward R, Edwards ST, Stange KC, Cohen DJ, Balasubramanian BA. Cardiovascular Disease Preventive Services Among Smaller Primary Care Practices. Am J Prev Med. 2022 May;62(5):e285-e295. doi: 10.1016/j.amepre.2021.10.011. Epub 2021 Dec 20. PMID 34937670
- [Result] Cohen DJ, Balasubramanian BA, Lindner S, Miller WL, Sweeney SM, Hall JD, Ward R, Marino M, Springer R, McConnell KJ, Hemler JR, Ono SS, Ezekiel-Herrera D, Baron A, Crabtree BF, Solberg LI. How Does Prior Experience Pay Off in Large-Scale Quality Improvement Initiatives? J Am Board Fam Med. 2022 Dec 23;35(6):1115-1127. doi: 10.3122/jabfm.2022.220088R1. PMID 36564196
- [Result] Sweeney SM, Baron A, Hall JD, Ezekiel-Herrera D, Springer R, Ward RL, Marino M, Balasubramanian BA, Cohen DJ. Effective Facilitator Strategies for Supporting Primary Care Practice Change: A Mixed Methods Study. Ann Fam Med. 2022 Sep-Oct;20(5):414-422. doi: 10.1370/afm.2847. PMID 36228060
- See also: National evaluation's public-facing website — http://escalates.org